CLINICAL TRIAL: NCT02012725
Title: Molecular MRI of the Fibrotic Heart
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Moriel Vandsburger (Other)
Responsible Party: Sponsor-Investigator, Moriel Vandsburger, Sponsor PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 5KL2TR000116-03 (NIH)
Record Dates: First submitted 2013-12-06; First posted 2013-12-16 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Healthy; Myocardial Fibrosis; Chronic Kidney Disease
Keywords: Healthy; Myocardial fibrosis; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Gadolinium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1 Mycardial Fibrosis: MRI with Intravenous administration of gadolinium
  Interventions: Drug: Arm 1 MRI with gadolinium
- Arm 2 Chronic Kidney Disease: MRI with no gadolinium administration

INTERVENTIONS:
Drug: Arm 1 MRI with gadolinium — Healthy volunteers will not receive gadolinium
  Groups: Arm 1 Mycardial Fibrosis

SUMMARY:
This study is a feasibility study to validate magnetizatin transfer (MT)-weighted balanced steady state free precession (bSSFP) cine cardiac magnetic resonance (CMR) against current clinical gold standard diagnostics, and to determine the applicability of MT-weighted bSSFP cine CMR for diagnosis of fibrotic remodeling in chronic kidney disease (CKD5) patients. Participants will not receive a study drug or placebo and will not be randomized. A total of 250 participants will be enrolled into this study.

DETAILED DESCRIPTION:
This study had two treatment arms.

Arm 1: Participants will be enrolled in this arm if they have been referred to the Gill Heart Institute MRI center for diagnostic late gadolinium enhancement (LGE) -CMR imaging of fibrosis, or if they are a healthy volunteer.

If a participant is a Gill Heart Institute referral patient , they will receive an intravenous (through a vein in the arm) infusion of gadolinium as part of their clinical examination. Participants will also have electrocardiogram (ECG) waveform performed in order to gate the MRI scan. The MRI scan of the heart, for which the participant has been referred will last approximately 1 hour. Participants will have an additional 5-10 minutes of scans performed, none of which require additional infusions.

If the participant is a healthy volunteer, they will have an ECG waveform performed in order to gate your MRI scan, and they will have approximately 30-45 minutes of scanning performed on their heart. Participants will not receive an infusion of gadolinium.

Arm 2: Only participants who are already participating in a study being conducted by Dr. Harmut Malluche at the University of Kentucky, Department of Nephrology or, if you are a healthy volunteer, will be enrolled into this arm.

In this arm participants will receive an MRI of their heart, lasting 30-45 minutes. Participants will not receive an infusion of gadolinium.

ELIGIBILITY:
Arm 1

Inclusion Criteria:

* Participants between the ages of 20 and 80
* Diagnosis or suspicion of myocardial fibrosis
* Referral for LGE-CMR

Exclusion Criteria:

* Confirmed acute MI within the prior 72 hours
* Unstable ECG or arrhythmia as determined by the referring physician
* Inability to hold one's breath for at least 10 seconds
* Standard MRI safety exclusion criteria
* Allergic reaction to Gadolinium
* Women who are pregnant, think they are pregnant or who breastfeeding

Arm 2

Inclusion Criteria:

* Participants between the ages of 20 and 80
* History of between 1-10 years of routine hemodialysis
* Healthy Volunteers

Exclusion:

* Confirmed acute myocardial infarction within the prior 72 hours
* Unstable ECG or arrhythmia
* Inability to hold one's breath for at least 10 seconds
* Standard MRI safety exclusion criteria

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants taking part in this study will be:
  * Referred from the University of Kentucky Gill Heart Institute (planned enrollment for this group is 100 patients)
  * Referred from another study on chronic kidney disease (planned enrollment for this group is 100 patients and 50 healthy volunteers)
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Arm 1 - Validation of gadolinium free fibrosis imaging against current standard of care LGE-CMR | 36 months
  Results from this arm will focus on validating cine FI measured from MT-weighted bSSFP cine CMR against LGE-CMR and MOLLI characterization of fibrosis in patients referred to the Gill Heart Institute.
Arm 2 - Imaging of myocardial fibrosis in CKD patients | 48 months
  Will test the hypothesis that MT-weighted CMR can be applied to identify fibrotic remodeling in the hearts of CKD5 patients

CONTACTS AND LOCATIONS:
Overall Officials: Moriel Vandsburger, PhD, Principal Investigator — University of Kentucky, Department of Physiology
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States